CLINICAL TRIAL: NCT00386321
Title: Yt90Zevalin Plus CHOP, Z-CHOP
Brief Title: Yt90 Zevalin and Combination Chemotherapy (Z-CHOP)in Treating Patients With Stage II, Stage III, or Stage IV Diffuse Large B-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Participants are no longer being examined or treated.
Sponsor: Chulalongkorn University (Other)
Collaborators: Bayer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH011103
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Zevalin; Zevalin plus CHOP; Diffuse large B-cell lymphoma; First line Diffuse large B-cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Yttrium 90 -labeled ibritumomab tiuxetan (Zevalin)

SUMMARY:
The purpose of this study is to determine whether the treatment of Yt90 Zevalin in combination with CHOP (cyclophosphamide, doxorubicin, vincristine, and prednisolone)are effective as first line treatment in patients with bulky stage II or stage III or IV diffuse large B-cell lymphoma

DETAILED DESCRIPTION:
Radioimmunotherapy represents a significant advance over unlabeled immunotherapy for the treatment of patients with B-cell non-Hodgkin's lymphoma. The radiobiological effects associated with Yt90-labelled ibritumomab tiuxetan (Zevalin) include the induction of apoptosis and cell-cycle redistribution.

The response rate tend to be higher in patients who have been treated with fewer prior therapies and Yt90-labelled ibritumomab tiuxetan may be suitable for use early in the course of therapy.

Yt90-labelled ibritumomab tiuxetan has less non hematologic toxicity than chemotherapy, with only minimal alopecia, mucositis, nausea, or vomiting, and a lower incidence of infections.

Yt90-labelled ibritumomab tiuxetan regimen is routinely and safely given in an outpatient setting and is completed in 7-9 days and is thus more convenient to be used.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20 positive diffuse large B-cell lymphoma with bulky stage II or stage III or stage IV
* Bidimensionally measurable disease
* Performance status Zubrod 0-2
* Less than 20,000/mcL circulating lymphoid cells on WBC differential count
* No clinical evidence of CNS involvement, no prior diagnosis of indolent lymphoma, no histologic transformation
* Ejection fraction more than or equal to 45% by MUGA or no significant abnormality by echocardiogram
* Fertile patients with effective contraception method
* No other malignancy within past 5 years except adequately treated basal cell or squamous cell skin cancer, stage I or II cancer in complete remission, or carcinoma in situ of cervix
* No HIV positive, no prior solid organ transplantation
* No prior antibody therapy, chemotherapy, radiotherapy for lymphoma

Exclusion Criteria:

* Serum creatinine ot bilirubin more than 2.5 X ULN unless due to lymphoma
* Active uncontrolled infection
* Concurrent severe and/or uncontrolled medical disease which could compromise participation in the study
* Patients with more than 25% infiltrated bone marrow
* Patients with platelet counts less than 100,000/mcL or neutrophil counts less than 1,500/mcL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-04; Primary Completion 2007-07 (Actual); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival and overall survival of patients

SECONDARY OUTCOMES:
Response rate (partial response, complete unconfirmed response, and complete response)in patients
2-year progression-free survival, overall survival and response rate in BCL-2 positive patients

CONTACTS AND LOCATIONS:
Overall Officials: Udomsak Bunworasate, M.D., Principal Investigator — Division of Hematology and Stem Cell Transplant, Department of Medicine, Faculty of Medicine, Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand